CLINICAL TRIAL: NCT05247632
Title: Precision Nutrition and Food Safety for Dietary Prevention of Chronic Disease (PNFS) Study
Brief Title: Precision Nutrition and Food Safety for Dietary Prevention of Chronic Disease Study
Acronym: PNFS
Status: Active, not recruiting | Type: Observational
Sponsor: Zhejiang University (Other)
Collaborators: Lanxi Red Cross Hospital (Unknown); Lanxi Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Yu Zhang, Professor, Zhejiang University
Other Study IDs: Cohort-PNFS
Record Dates: First submitted 2022-02-03; First posted 2022-02-21 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2023-03

CONDITIONS: Chronic Diseases
Keywords: Food safety; Food nutrition; Food contaminant; Mult-omics; Chronic diseases
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The investigators collected blood samples.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The associations between food nutrition and safety factors with the risk of chronic diseases are still unclear. This study is conducted in Jinhua, a city with a high prevalence of chronic diseases in China, to assess relations between food nutrition and safety factors and chronic diseases.

DETAILED DESCRIPTION:
Investigations of associations of food nutrition and safety factors with the risk of chronic diseases are limited and studies in China are still lacking. The investigators aim to collect basic characteristics of participants at baseline, including sex, age, smoking, exercise, marriage, education level, dietary factors, and so on, to assess the association of food nutrition and safety factors including various food items, dietary fatty acids, and internal biomarkers of food contaminants such as acrylamide and 3-MCPD with various chronic diseases in a Chinese middle-aged and elderly population. We will use multi-omics technology to investigate the causal mechanisms. Results from this study will be valuable for chronic diseases prevention in China.

ELIGIBILITY:
Inclusion Criteria:

* Subject aged ≥45 and ≤74 years old
* Subject has complete data on diet and follow-up time

Exclusion Criteria:

had the major illness that had made personal life disabled

Ages: 45 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects are eligible residents from 10 government-administered units including 7 urban towns and 3 rural villages of Jinhua, China.
Sampling Method: Probability Sample
Enrollment: 2290 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Numbers of participants with metabolic syndrome | From entry into the study baseline:2018 until 2023
  metabolic syndrome
Numbers of participants with obesity | From entry into the study baseline:2018 until 2023
  Obesity
Numbers of participants with diabetes | From entry into the study baseline:2018 until 2023
  Diabetes

SECONDARY OUTCOMES:
Numbers of participants died | From entry into the study baseline:2018 until 2023
  All-cause and cause-specific mortality
Numbers of participants with cardiovascular diseases | From entry into the study baseline:2018 until 2023
  Cardiovascular diseases

OTHER OUTCOMES:
Numbers of participants with fatty liver disease | From entry into the study baseline:2018 until 2023
  Fatty liver disease

CONTACTS AND LOCATIONS:
Overall Officials: Weifang Zheng, Study Director — Lanxi Red Cross Hospital; Jingjing Jiao, Principal Investigator — Zhejiang University; Yu Zhang, Principal Investigator — Zhejiang University; Pan Zhuang, Principal Investigator — Zhejiang University
Locations (2):
- China (2):
  - Lanxi Red Cross Hospital, Lanxi, Zhejiang
  - Lanxi Hospital of Traditional Chinese Medicine, Jinhua